CLINICAL TRIAL: NCT03566524
Title: Arginine and Nitric Oxide Synthesis in the Pathogenesis of Ketosis-prone Diabetes
Brief Title: Study of Arginine and Nitric Oxide in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Farook Jahoor, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DK101411
Record Dates: First submitted 2018-05-31; First posted 2018-06-25 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Ketosis Prone Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Citrulline; Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citrulline (Experimental): In this arm, 10 ketosis prone diabetes patients will be randomly assigned to receive 34.2 mmol/d of dietary citrulline for 20 days. Citrulline will be in the form of 2.85 mmol capsules and patients will be instructed to consume 4 capsules with each of their 3 main meals. The citrulline will be provided in a double-blind fashion by a designated unblinded investigator who will not come in direct contact with the subjects.
  Interventions: Dietary Supplement: Citrulline
- alanine (Placebo Comparator): In this arm, 10 ketosis prone diabetes patients will be randomly assigned to receive 34.2 mmol/d of dietary alanine for 20 days. Alanine will be in the form of 2.85 mmol capsules and patients will be instructed to consume 4 capsules with each of their 3 main meals. The alanine will be provided in a double-blind fashion by a designated unblinded investigator who will not come in direct contact with the subjects.
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Citrulline — Ketosis prone diabetes patients (n=10) will be randomly assigned to receive either dietary supplement of citrulline or alanine as placebo. They will then cross over to the other supplement.
  Arms: Citrulline
Dietary Supplement: Alanine — Ketosis prone diabetes patients (n=10) will be randomly assigned to receive either dietary supplement of citrulline or alanine as placebo. They will then cross over to the other supplement.
  Arms: alanine

SUMMARY:
This study will test the effect of citrulline versus placebo supplementation in ketosis-prone diabetes (KPD) patients on arginine and nitric oxide production and on glucose- and arginine-stimulated insulin secretion and arterial flow-mediated dilation.

DETAILED DESCRIPTION:
Both arginine and its derivative nitric oxide (NO) have been implicated in the regulation of glucose homeostasis. Arginine is a β cell secretagogue, potentiating glucose stimulated insulin secretion. Further, it has been shown that glucose can stimulate NO production in primary β cells, and NO then enhances insulin secretion.

On the other hand, because the only known fate of citrulline is its conversion to arginine, citrulline supplementation could be a more efficient and safe way to increase intracellular arginine. Compared to enteral arginine, citrulline administration to healthy humans elicited a greater increase in plasma arginine and NO products, suggesting a greater increase in cellular arginine availability for NO synthesis. Therefore dietary citrulline supplementation will result in greater arginine availability and NO synthesis than arginine supplementation per se in KPD patients. In addition, because the consequences of diminished NO production in usual type 2 diabetes includes vascular dysfunction, an overall increase in NO production in response to citrulline supplementation will result in an improvement in vascular function assessed by arterial flow-mediated dilation

ELIGIBILITY:
Inclusion Criteria:

* New onset (defined as receiving a diagnosis within the past 1 year) diagnosis of unprovoked" A-β+ ketosis-prone diabetes
* Aged 20-65 years
* In good health except for diabetes without clinical evidence of micro- or macrovascular complications by history, physical exam and blood chemistries

Exclusion Criteria:

* Chronic or acute illness
* History of myocardial infarction or coronary artery disease or stroke,
* Renal insufficiency (eGFR <90mL/min/1.73m2; <30 mg albumin / g creatinine in urine)
* Abnormal liver, thyroid, gonadal or adrenal functions
* On medications other than metformin,
* On any hormonal replacement therapy
* Pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Arginine production | Three weeks
  The change in the amount of arginine produced from baseline in response to supplements of citrulline versus alanine (placebo) will be assessed by stable isotope tracers after 3 weeks of supplementation.

SECONDARY OUTCOMES:
Change in Nitric Oxide Synthesis | Three weeks
  The change in the amount of nitric oxide produced produced from baseline in response to supplements of citrulline versus alanine (placebo) will be assessed by stable isotope tracers after 3 weeks of supplementation.
Change in Arterial function | Three weeks
  The change in in arterial function (assessed by endopat) from baseline in response to supplements of citrulline versus alanine placebo will be assessed after 3 weeks of supplementation.
Change in Insulin secretion | Three weeks
  The change in glucose stimulated insulin secretion from baseline in response to supplements of citrulline versus alanine placebo will be assessed after 3 weeks of supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor St Lukes Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No